CLINICAL TRIAL: NCT00186537
Title: Comparison Fenofibrate, Rosiglitazone, or Weight Loss to Decrease Cardiovascular Risk in Insulin Resistant Dyslipidemic Individuals.
Brief Title: Comparing Tricor, Avandia, or Weight Loss to Lower Cardiovascular Risk Factors in People With High Triglycerides.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Gerald M Reaven, Professor Emeritus, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 79301; SPO 28829
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Insulin Resistance; Hypertriglyceridemia
Keywords: Insulin resistance; Insulin resistance syndrome; dyslipidemia; atherogenic dyslipidemia; triglyceride/HDL-C ratio
MeSH Terms: conditions — Insulin Resistance; Hypertriglyceridemia; Metabolic Syndrome; Dyslipidemias | interventions — Rosiglitazone; Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- fenofibrate (Active Comparator): 160 mg daily for 12 weeks
  Interventions: Drug: Fenofibrate
- rosiglitazone (Active Comparator): 4 mg/daily 4 weeks followed by 4 mg 2 x daily for 8 weeks
  Interventions: Drug: Rosiglitazone
- calorie restricted diet (Active Comparator): calorie restricted to achieve 0.5 kg weight loss/week x 12 weeks
  Interventions: Behavioral: Weight Loss

INTERVENTIONS:
Drug: Rosiglitazone
  Other Names: avandia
  Arms: rosiglitazone
Drug: Fenofibrate
  Other Names: tricor
  Arms: fenofibrate
Behavioral: Weight Loss
  Arms: calorie restricted diet

SUMMARY:
Approximately 1/4 of the US population has insulin resistance and the associated risk factors such as elevated lipid levels -triglycerides (type of fat from what we eat and what the liver produces and low HDL cholesterol which is the good cholesterol helping to protect against heart disease. Currently one known treatment for this a medication called fenofibrate, another medication that can improve insulin resistance is rosiglitazone, a third treatment known to improve insulin resistance an decrease triglycerides is weight loss. In this study insulin resistant individuals with elevated triglycerides and or a ratio of triglycerides to HDL cholesterol of 3:1 or greater will be randomized (selected by chance) to receive one of these treatments and results of insulin sensitivity and cardiac risk profiles will be compared at the end of the study.

DETAILED DESCRIPTION:
It has been estimated that approximately ¼ of the US population has the Insulin Resistant Syndrome (IRS). The notion that insulin resistance and compensatory hyperinsulinemia lead to a cluster of abnormalities that increase CVD risk was first introduced in 1988, and central to the changes identified was a dyslipidemia characterized by a high plasma triglyceride (TG) and low high-density lipoprotein cholesterol (HDL-C) concentration. The atherogenic lipoprotein pattern associated with the IRS has grown to include enhanced postprandial lipemia and smaller and denser low-density lipoprotein (LDL) particles. In addition to being associated with insulin resistance and compensatory hyperinsulinemia, these changes in lipoprotein metabolism have been identified as increasing CVD risk. The power of the dyslipidemia associated with the IRS is reinforced by reports that the plasma TG/HDL-C concentration ratio is as powerful a predictor of CVD, if not more so, than the more conventional total plasma cholesterol/LDL-C concentration ratio, and evidence from the Copenhagen Male Study of the interaction between the plasma TG and HDL-C concentrations, "conventional" CVD risk factors, and CVD events. Specifically, these latter investigators were able to show in a prospective study (11) that CVD events were substantially attenuated in: 1) smokers; 2) patients with high blood pressure; 3) individuals with a high LDL-C concentration; and 4) subjects who were sedentary; as long as they were in the lowest 1/3rd of the population with the lowest TG/HDL-C concentration ratio and presumably insulin sensitive. Conversely, if they were in the tertile with the highest plasma TG/HDL-C concentration ratio, and presumably insulin resistant, they had a significant increase in CVD events in the absence of the four conventional CVD risk factors evaluated.

An obvious alternative therapeutic approach to decreasing CVD risk in patients with the IRS would be to administer a thiazolidinedione (TZD) compound in an effort to directly treat the basic defect of the syndrome. However, based upon our own results with rosiglitazone (ROSI) in several different patient populations, improvements in insulin sensitivity were not associated with a significant improvement in dyslipidemia. For example, in a recent study (unpublished) of ROSI-treated patients with type 2 diabetes, neither plasma TG (358 to 347 mg/dL) nor HDL-C (40 to 42 mg/dL) concentrations improved, and both total (215 to 239 mg/dL and LDL-C (118-142mg/dL) concentrations actually increased. Since the patients in this study became more insulin sensitive with treatment, and had lower daylong plasma glucose, insulin, and free fatty acid concentrations, the reason for the lack of a beneficial effect of ROSI on lipoprotein metabolism is not clear. On the other hand, given evidence of the importance of dyslipidemia in increasing CVD risk in insulin resistant individuals, it seems reasonable to question the notion that TZD compounds provide the most beneficial approach to decreasing CVD risk in the dyslipidemic patient with the IRS.

With this background in mind, we propose to initiate a study in which insulin resistant individuals with the dyslipidemia characteristic of the IRS will be randomized to treatment with fenofibrate,ROSI, or weight loss and the effect of these three treatments on CVD risk factors compared. It is postulated that although insulin resistance will improve to a greater degree with ROSI treatment, the atherogenic lipoprotein profile known to link IRS and CVD will only significantly improve following treatment with fenofibrate and effects of weight loss can effect both of these.

ELIGIBILITY:
Inclusion Criteria:

Insulin Resistant Triglyceride 150 mg/dL or greater or triglyceride HDL-C ratio 3 or greater BMI 25-35

Exclusion Criteria:

Diabetes Mellitus History of gall stones History of CHF History of CAD Severe anemia,kidney, or liver disease

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2003-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald M Reaven, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reaven GM. Banting lecture 1988. Role of insulin resistance in human disease. Diabetes. 1988 Dec;37(12):1595-607. doi: 10.2337/diab.37.12.1595. PMID 3056758
- [Background] Laws A, Reaven GM. Evidence for an independent relationship between insulin resistance and fasting plasma HDL-cholesterol, triglyceride and insulin concentrations. J Intern Med. 1992 Jan;231(1):25-30. doi: 10.1111/j.1365-2796.1992.tb00494.x. PMID 1732395
- [Background] Ford ES, Giles WH, Dietz WH. Prevalence of the metabolic syndrome among US adults: findings from the third National Health and Nutrition Examination Survey. JAMA. 2002 Jan 16;287(3):356-9. doi: 10.1001/jama.287.3.356. PMID 11790215

RESULTS

PARTICIPANT FLOW:
Groups:
- Fenofibrate: 160 mg daily for 12 weeks
  Fenofibrate
- Rosiglitazone: 4 mg/daily 4 weeks followed by 4 mg 2 x daily for 8 weeks
  Rosiglitazone
- Calorie Restricted Diet: calorie restricted to achieve 0.5 kg weight loss/week x 12 weeks
  Weight Loss
Period: Overall Study
Arm/Group | Fenofibrate | Rosiglitazone | Calorie Restricted Diet
Started | 19 | 12 | 16
Completed | 12 | 12 | 13
Not Completed | 7 | 0 | 3
Not completed — Withdrawal by Subject | 4 | 0 | 3
Not completed — ALT > 1.5 x ULN | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis was done on those who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Fenofibrate | Rosiglitazone | Calorie Restricted Diet | Total
Number analyzed (Participants) | 12 | 12 | 13 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7) | 52 (6) | 53 (7) | 53 (7)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 5 | 6 | 14
  Male | 9 | 7 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Pre- and Post-Intervention Triglyceride Levels
Description: Compare the change in mean triglyceride levels between groups after the interventions
Time Frame: Baseline, 12 weeks
Population: Triglycerides
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fenofibrate | Rosiglitazone | Calorie Restricted Diet
Number analyzed (Participants) | 12 | 12 | 13
mg/dL
  pre treatment | 231 (117) | 209 (67) | 201 (121)
  post treatment | 140 (47) | 232 (72) | 143 (49)

2. Primary Outcome: Pre- and Post-Intervention LDL Cholesterol Levels
Description: Compare the change in mean LDL Cholesterol levels between groups after the interventions
Time Frame: Baseline, 12 weeks
Population: LDL cholesterol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fenofibrate | Rosiglitazone | Calorie Restricted Diet
Number analyzed (Participants) | 12 | 12 | 13
mg/dL
  pre treatment | 114 (34) | 119 (41) | 144 (34)
  post treatment | 111 (22) | 129 (37) | 128 (34)

3. Primary Outcome: Pre- and Post-Intervention HDL Cholesterol Levels
Description: Compare the change in mean HDL Cholesterol levels between groups after the interventions
Time Frame: Baseline, 12 weeks
Population: HDL Cholesterol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fenofibrate | Rosiglitazone | Calorie Restricted Diet
Number analyzed (Participants) | 12 | 12 | 13
mg/dL
  pre treatment | 35 (7) | 40 (11) | 38 (9)
  Post treatment | 36 (8) | 42 (13) | 38 (7)

ADVERSE EVENTS:
Arm/Group | Fenofibrate | Rosiglitazone | Calorie Restricted Diet
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/12 | 0/16
Other Adverse Events (participants affected / at risk) | 3/19 | 0/12 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate (N=19) | Rosiglitazone (N=12) | Calorie Restricted Diet (N=16)
alanine aminotramsferase ( ALT) elevation greater than 1.5 times normal of upper limit (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes